CLINICAL TRIAL: NCT03896555
Title: Intrafractional 6D Head Movement With Mask Fixation During Stereotactic Intracranial RT-sessions
Brief Title: Intrafractional Head Movement During Radiosurgery
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: intrafractpos_2019
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-01

CONDITIONS: Brain Metastases, Adult
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ExacTrac position verification — Repeated measurement of patient head position with ExacTrac X-ray Monitoring

SUMMARY:
This study investigates the intrafractional accuracy of a frameless thermoplastic mask used for head immobilization during stereotactic radiotherapy. Non-invasive masks cannot completely prohibit head movements. Previous studies attempted to estimate the magnitude of intrafractional inaccuracy by means of pre- and postfractional measurements only. However, this might not be sufficient to accurately map also intrafractional head movements.

Intrafractional deviation of mask-fixed head positions is measured in five patients during a total of 94 fractions by means of close-meshed repeated ExacTrac measurements conducted during the entire treatment session. From the obtained data the investigators evaluate the need to adjust safety margins around the gross tumor volume (GTV) whenever the investigated thermoplastic mask is used instead of invasive ring fixation.

ELIGIBILITY:
Inclusion Criteria:

* single intracranial tumour or metastasis
* stereotactic radiation therapy planned
* immobilization with thermoplastic mask

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 5 Patients with a single intracranial tumour treated with stereotactic radiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
3D Head deviation | 5 to 20 days
  Length of 3D head position deviation during RT session

CONTACTS AND LOCATIONS:
Overall Officials: Meinhard Nevinny-Stickel, MD, PhD, Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: Yes
De-identified Datasets of all measured parameters will be made available
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after publication
Access Criteria: The datasets used and analysed during the study will be available from the corresponding author on reasonable request

REFERENCES:
- [Derived] Mangesius J, Seppi T, Weigel R, Arnold CR, Vasiljevic D, Goebel G, Lukas P, Ganswindt U, Nevinny-Stickel M. Intrafractional 6D head movement increases with time of mask fixation during stereotactic intracranial RT-sessions. Radiat Oncol. 2019 Dec 18;14(1):231. doi: 10.1186/s13014-019-1425-7. PMID 31852497

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT03896555/Prot_SAP_000.pdf